CLINICAL TRIAL: NCT03952676
Title: Clinical Evaluation of Moving Cupping for Plaque Psoriasis: a Randomized Controlled Trial
Brief Title: Moving Cupping for Plaque Psoriasis: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Shaanxi Traditional Chinese Medicine Hospital (Unknown); Heilongjiang University of Chinese Medicine (Other); Shijiazhuang traditional Chinese medicine hospital (Unknown); The Affiliated Hospital of JiangXi University of TCM (Unknown); Xinjiang Uygur Autonomous Region Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018YFC1705303
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis; Blood stasis syndrome; Randomized controlled trial; Moving cupping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moving cupping intervention (Experimental): Participants will received moving cupping therapy once a week for 4 weeks.In addition, participants will receive basic treatment, including the use of moisturizing lotion, avoid induction and aggravating factors, proper bathing to clean the skin, reasonable lifestyle and treatment.
  Interventions: Device: Moving cupping
- Moving cupping placebo control (Placebo Comparator): Participants will received moving cupping placebo therapy once a week for 4 weeks.In addition, participants will receive basic treatment, including the use of moisturizing lotion, avoid induction and aggravating factors, proper bathing to clean the skin, reasonable lifestyle and treatment.
  Interventions: Device: Moving cupping placebo

INTERVENTIONS:
Device: Moving cupping — 1. We use a black opaque eye mask to shield the patient's eyes and choose different sizes of cup according to the location of the treatment (There are three sizes of cups)
  2. (1) First apply Vaseline to the skin lesions area; (2) Then hold the 95% ethanol cotton ball with tweezers, and hold the cup with the facing down, after the cotton ball is ignited, immediately sway down in the cup and then exit, and quickly buckle the cup to the skin lesions area. (3) After using the cup to absorb the skin lesions area, hold the cup body in one hand and push and pull the cup along the certain route with a little strength, so that the skin purple color of the treatment area is suitable. (4) Apply even force when pushing the cup to prevent the cup from falling off due to air leakage. (5) Acting on the skin lesions area 30 times, change cup 5 times per push and pull, the interval is not more than 10 seconds.
  Arms: Moving cupping intervention
Device: Moving cupping placebo — Using of special perforated cups, the manipulation method is the same as the intervention group.
  Arms: Moving cupping placebo control

SUMMARY:
The purpose of this study was to provide evidence support for the effectiveness and safety of moving cupping therapy for plaque psoriasis through clinical studies.

DETAILED DESCRIPTION:
Psoriasis is a common chronic and recurrent inflammatory skin disease. The incidence of the disease is increasing year by year, seriously affecting people's quality of life. The systematic treatment of psoriasis in modern medicine is limited of wide application due to the adverse reactions of different degrees and the high economic cost.

Complementary and alternative medicine (CAM) therapies have become an increasingly visible part of dermatology. Cupping is becoming an important therapy in complementary and alternative medicine. Although, moving cupping therapy has been widely used in the treatment of plaque psoriasis and has been recognized by a large number of peers and patients, but still lacks high-quality evidence-based medical evidence. Therefore, the project team intends to provide evidence support for the effectiveness and safety of moving cupping therapy for plaque psoriasis through clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic criteria for plaque psoriasis;
2. Skin lesions involve ≤10% BSA (the lesions are mainly located in the torso / limbs, palm / sole, face / scalp, vulva area is not included);
3. Aged between 18 and 65 years.
4. Consent to participate in the research study and sign the informed consent form

Exclusion Criteria:

1. Patients with pustular psoriasis, arthropathic, erythroderma psoriasis and / or drip psoriasis;
2. Plaque psoriasis patients with BSA>10%;
3. Any clinically active skin diseases other than moderate to severe psoriasis vulgaris which might counter or influence the study aim;
4. Patients who used any of the following systemic treatments within 4 weeks before the Baseline visit e.g.: drugs for other studies, immuno-suppressive drugs, biologics;
5. Patients who used topical treatment within 2 weeks before the Baseline visit e.g. corticosteroids ultraviolet-light therapy including sunbathing;
6. Active infectious disease which was hard to control;
7. History of severe systemic disease. Or the clinical test index is one of the following: the ALT or the AST is higher than 1.5 times; Any of the main routine blood indexes (WBC, RBC, HB, PLT) is lower than the limit of normal; or other laboratory abnormalities and patients were judged not to be suitable for this study;
8. Family history of cancer-prone patients;
9. Patients with immunocompromised and can cause skin allergies and infection when moving cupping;
10. Pregnant or lactating women;
11. Patients with a history of alcohol abuse and drug abuse;
12. Have a history of serious mental illness or family history; 13 Other reasons researchers believe that patients are not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Psoriasis area and severity index (PASI) | Up to 56 days after treatment
  Psoriasis Area and Severity Index (PASI) involves grading psoriatic plaques based on erythema (E), infiltration (I), desquamation (D). Severity is graded from 0-4 for each criteria (0 - none, 1 - slight, 2 - moderate, 3 - severe, and 4 - very severe). The body is divided into 4 regions, head, upper extremities, trunk, and lower extremities, and for each region, the surface area involvement is graded on a 0-6 scale (0 - 0% involvement, 1 - <10%, 2 - 10-<30%, 3 - 30-<50%, 4 - 50-<70%, 5 - 70-<90%, 6 - 90-100%).The highest potential PASI score is 72, with higher PASI scores indicating worse psoriasis.

SECONDARY OUTCOMES:
Body surface area (BSA) | Up to 56 days after treatment
  The percentage of BSA involved in psoriasis is estimated by fingerprinting, where the entire palm of the patient represents approximately 1% of the total BSA. The number of handprints on psoriasis skin in a body part is used to determine the extent to which the body part is affected by psoriasis (%).
Physician Global Assessment (PGA) | Up to 56 days after treatment
  Physician Global Assessment (PGA) is scored on a 5-point scale, reflecting a global consideration of the erythema (E), infiltration (I), desquamation (D) across all psoriatic lesions. It is calculated as follows: PGA score = (E + I + D) / 3, then the score needs to be rounded to the nearest whole number [PGA scale: Clear (0) - Very Severe (5)].
Dermatology Life quality index(DLQI) | Up to 28 days after treatment
  The Dermatology Life Quality Index (DLQI) is a participant-reported questionnaire used to measure the health-related quality of life (QOL) of adults suffering from a skin disease. Scores range from 0-30, a higher score indicating a greater impact on a participant's quality of life.
Patient-reported quality of life (PRQoL) | Up to 28 days after treatment
  PRQoL is used to assess the impact of psoriasis on individual social life. Scores range from 0-25, a higher score indicating a greater impact on a participant's social life.
Visual Analogue Score (VAS) | Up to 56 days after treatment
  Visual Analog Scale (VAS) is used to measure lesion pruritus from 0 to 100 mm at eash visit (with 0 being no pruritis and 100 being maximum pruritis).
CM symptom score | Up to 28 days after treatment
  The CM symptom score is used to assess changes in blood syndrome related symptoms during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, Study Chair — Shanghai Yueyang Integrated Medicine Hospital
Locations (5):
- China (5):
  - First Affiliated Hospital, Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - The Affiliated Hospital of Jiangxi University of TCM, Nanchang, Jiangxi
  - Shaanxi Provincial Hospital of traditional Chinese Medicine, Xi'an, Shaanxi
  - Shijiazhuang traditional Chinese medicine hospital, Shijiazhuang, Shijiazhuang
  - Xinjiang Uygur Autonomous Region Traditional Chinese Medicine Hospital, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xing M, Yan X, Yang S, Li L, Gong L, Liu H, Xu R, Chen J, Ying L, Zhao Y, An Y, Liu Y, Huang G, Guo F, Yin Q, Wang R, Li B, Li X. Effects of moving cupping therapy for plaque psoriasis: study protocol for a randomized multicenter clinical trial. Trials. 2020 Feb 26;21(1):229. doi: 10.1186/s13063-020-4155-0. PMID 32102679